CLINICAL TRIAL: NCT05806593
Title: Get Back, a Person-centred Digital Program Targeting Physical Activity for Patients Undergoing Spinal Stenosis Surgery - a Randomized Feasibility Study
Brief Title: Feasibility of a Person-centred Digital Program Targeting Physical Activity in Spinal Stenosis Surgery
Acronym: GetBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophiahemmet University (Other)
Collaborators: The Swedish Research Council (Other Government); AFA Insurance (Industry)
Responsible Party: Principal Investigator, Mari Lundberg, Professor, Sophiahemmet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Get Back
Record Dates: First submitted 2023-03-11; First posted 2023-04-10 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Spinal Stenosis Lumbar
Keywords: Health promotion; Person-centred care; Physical activity; Behavioral medicine; Telehealth
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Get Back pilot) (Experimental): The intervention includes 5 core sessions (video call) and 5 booster sessions (telephone) over 12 weeks (1 week before until 11 weeks after surgery). All sessions will be led by a physiotherapist. The focus of each core session (1-5) is as follows:
  1. To establish the patient as an active, equal partner in the treatment and to formulate a shared health plan according to person-centred care.
  2. To reduce the threat value of postoperative pain and increase the patient's knowledge about the biopsychosocial nature of pain and positive effects of physical activity.
  3. To detect barriers for postoperative physical activity and to support the patient to gradually start increasing physical activity.
  4. To increase approach behavior for physical activity and reduce avoidance behavior by confronting fears and move towards personal goals.
  5. To support the patient to independently continue with activity progress towards long term health and to formulate a maintenance plan.
  Interventions: Behavioral: Get Back pilot
- Control (standard physiotherapy) (No Intervention): The control group will follow standard physical therapy, meaning physical therapy as it is provided at each recruiting site when undergoing surgery due to spinal stenosis. As this may differ substantially between clinical sites nationally, data on frequency of physical therapy and the content of the physical therapy sessions during the study period will be collected as a control variable weekly from the control group.

INTERVENTIONS:
Behavioral: Get Back pilot — A health-promoting program, targeting physical activity behavior, with a person-centred approach led by a physiotherapist digitally during 12 weeks.
  Arms: Intervention (Get Back pilot)

SUMMARY:
Spinal stenosis is the most common cause of degenerative spinal surgery. The majority do not achieve the global recommendations for health-promoting physical activity before or after surgery. Patients with a low level of physical activity and a high degree of fear of movement are at an increased risk of poorer health outcomes after surgery. Increasing the number of steps per day is a way to increase physical activity, which in long term can lead to health benefits. In addition, a digital format is a way to increase the availability of physiotherapy to strive for equal rehabilitation.

The overall purpose of the research project is to improve health outcome and increase the availability of rehabilitation for patients at high risk of negative health outcomes after spinal surgery due to spinal stenosis through Get Back, a person-centered and digital program with a focus on physical activity.

Before conducting a large-scale study, the investigators want to conduct a study that aims to investigate and develop the Get Back program regarding content and dose, treatment fidelity as well as feasibility in terms of study procedure, compliance, and acceptability.

Approximately thirty patients with lumbar spinal stenosis and an identified risk profile for poorer postoperative outcomes will be recruited from two spine clinics in Sweden. The program involves meeting a physiotherapist digitally (through video call) approximately 1 week before surgery to formulate a person-centered health plan. The health plan is monitored and progressed by the physiotherapist by video until eleven weeks after surgery. The Get Back program includes 5 sessions (1 hour each) which are supplemented with 5 booster sessions (30 minutes) to reinforce the intervention. Get Back is based on three key components that run through all sessions. These are person-centeredness, behavioral medicine techniques to reduce fear of movement and worries about pain, as well as to optimize physical activity. The physiotherapist supports the participant's individual resources and abilities through validated behavioral medicine methods in combination with education/communication/knowledge support and behavior-strengthening tools (which are also used in-between sessions) to achieve the participant's personal goals linked to physical functioning, physical activity, and health. The program will be compared to standard physiotherapy.

DETAILED DESCRIPTION:
Get Back is developed based on a prior person-centered prehabilitation program for patients undergoing lumbar fusion surgery. The prior program showed good effect on the patient's health directly after the intervention, had a high adherence rate and was found to be safe. The prior program was, however, conducted on a relatively healthy and young group (age 46 years). Get Back aims to expand this program to include patients with lumbar spinal stenosis (LSS), who are at risk of negative health outcomes after surgery. Get Back will be delivered by e-health (video calls) as prior face-to-face interventions have identified barriers for participation by long travel distances to the rehabilitation centre. The program will focus on health promotion throughout the whole perioperative period in contrast to previous programs that have focused on reducing disability. Get Back will target for example walking behavior with the aim to increase the patients' physical activity (primarily assessed by steps per day as a proxy), as it is associated with a progressively lower risk of all-cause mortality. Before the investigators start a full scale randomized controlled trial, a feasibility trial will be conducted to assure and refine the evaluation design and the intervention, recommended by The Medical Research Council (MRC).

Participants will be recruited from two private spine clinics located in two different regions. Patients will be clinically examined by an orthopaedic surgeon, who will make a medical diagnosis based on the clinical and radiological findings. If a surgical decision is made and the patient is placed on the waiting list, a physiotherapist will contact the patient meeting inclusion criteria and screen for the risk profile as well as provide the information about the study and ask for participation. As the intervention is fully digital the patient information in written will also be sent to the patient digitally. Inclusion and exclusion criteria are described under paragraph 10.

The primary study aim is to explore if Get Back can provide a detectable change in variables related to the intervention content (steps per day, physical activity level, as well as variables related to pain catastrophizing, fear of movement, and self-efficacy) and to evaluate treatment fidelity as well as feasibility in terms of trial procedure, compliance, and acceptability. A randomized feasibility study (n=30) with multiple measures will be conducted in preparation for a future two-arm multicenter randomized controlled trial.

At baseline, approximately 2 weeks before surgery, all participants, will meet with an independent observer digitally (video call) who will collect demographic data, and conduct a few physical function tests. The patient will fill in patient reported outcome measures (PROMs) digitally. An accelerometer will be sent out to the study participant through mail to wear for 7 days. A study coordinator will then allocate the patients to either the Get Back pilot (n= 15) or standard physiotherapy (n= 15) based on a computerized random list converted to concealed envelopes. The independent observer will be blinded to group allocation. The assessment battery (demographic data will be replaced by clinical data) will be repeated at the end of the intervention (approx. 11-12 weeks after surgery). The intervention-group will also have an addition of a telephone based semi structured interview regarding feasibility aspects and participation. Each week during the intervention participants will digitally answer one-item questions based on the included PROMs, (described in detail under "data collection").

Get Back pilot includes five core session and will be led by the PT-Get Back. The core session will be complemented by up to five shorter follow ups by telephone (booster sessions). The intervention in described more in detail under paragraph 8.

Outcome measurements are described in detail under paragraph 9. Treatment fidelity data including intervention dose, content, and adherence to intervention procedures will be collected.

Process and resource feasibility will be administrated by the variables: recruitment, session compliance, safety, and acceptability.

Feasibility data will be collected continuously during and at the end of the study period.

Data from accelerometer, patient reported outcome measures and physical capacity tests will be collected at baseline, and 11-12 weeks after surgery. Baseline variables such as age, gender, comorbidity, ASA-score, weight/height, smoking status, alcohol consumption, educational level, sick-leave status, pain duration (back and leg), and previous spine surgery will be collected from the patient. Preoperative cognitive function will be measured with the Cognitive Performance Scale. Pre- and postoperative clinical data such as type of surgery, complications, length of stay, analgesic use, discharge destination, re-operation, and re-admission to hospital will be collected from the medical records at each recruiting unit. For the standard physiotherapy group, pre- and postoperative physical therapy will also be collected as a control variable. Weekly measures will include one-item questions including steps per day, physical activity level, as well as variables related to pain catastrophizing, fear of movement, and self-efficacy. Weekly measures will be conducted digitally and take approximately 5 minutes to fill in.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for decompression surgery (no fusion) due to central lumbar spinal stenosis
* reporting a low level of physical activity (do not meet WHO´s physical activity recommendations of minimum 150 min moderate intensity per week), and one of the following criteria at preoperative screening; fear of movement (Tampa Scale of Kinesiophobia (TSK) ≥ 37) and/or pain catastrophizing (Pain Catastrophizing Scale (PCS) >30).

Exclusion Criteria:

* Patients with malignancy, severe neurological -or rheumatic disease, idiopathic scoliosis, isthmic spondylolisthesis
* not able to understand written information and communicate in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Change in variables related to intervention content. | Once a week during the 12-week study period.
  A questionnaire including 14 one-item questions aiming to capture steps per day (reported from a pedometer), self-reported physical activity level, and relevant aspects of pain catastrophizing, fear of movement and self-efficacy (on rating scales ranging from 0 to 10).
The intervention participants frequency and length of contact with the study physiotherapist. | Continuously during the 12 week intervention.
  The data will be noted by the study physiotherapist on each session protocol.
Checklist of included components at each treatment session. | Continuously during the 12 week intervention.
  The treatment components addressed during each intervention session will be noted by the study physiotherapist on a checklist.
Analysis of audio recordings from the intervention sessions. | Continuously during the 12 week intervention.
  Audio recordings of the intervention sessions will be conducted and transcribed for post-hoc analysis by a third party (trained in person centredness and cognitive behavioural therapy) to ensure that the key components of the intervention are included.
Type and frequency of possible adverse events. | Continuously during the 12 week intervention.
  The type and frequency of possible adverse events during the intervention will be collected by the study physiotherapist and noted on each session protocol.
Percentage of patients eligible after the screening procedure. | Through study completion, an average of 6 month.
  The data will be noted on screeninglists.
Number of intervention sessions attended out of planned. | Through study completion for each intervention participant, an average of 12 weeks.
  The data will be noted by the study physiotherapist on each session protocol.
Acceptability of data collection methods measured with a study specific questionnaire. | At the end of each participants 12 week study period.
  Study specific questionnaires including questions related to experiences from participants and assessors of the methods used for data collection.
Participants experiences of the intervention collected via telephone interviews. | At the end of intervention/after 12 weeks.
  Semi structured telephone interviews with participants of the intervention group, which will be audio recorded and transcribed into text material.

SECONDARY OUTCOMES:
Steps per day collected with a activity tracker/accelerometer (Actigraph GT3X+). | At baseline, and post-intervention/after 12 weeks
  Reported as number of steps per day.
Physical activity level collected with a activity tracker/accelerometer (Actigraph GT3X+). | At baseline, and post-intervention/after 12 weeks
  Reported as time spent in light physical activity, moderate to vigorous physical activity (MVPA) and time spent sedentary.
Physical function measured with the Timed-up-and-go test (TUG). | At baseline, and post-intervention/after 12 weeks
  The time it takes for a participant to rise from a chair, walk 3 meters, turn, walk back to the chair and sit down. Reported in seconds.
Postural balance measured with the One Leg Stand test. | At baseline, and post-intervention/after 12 weeks
  The time a participant can stand on one leg, reported in seconds.
Functional leg strength measured with the 30 seconds sit-to-stand test. | At baseline, and post-intervention/after 12 weeks
  Reported as the number of chair rises a participant can complete during 30 seconds.
Self-reported physical activity collected with a two-item questionnaire from the National Board of Health and Welfare in Sweden. | At baseline, and post-intervention/after 12 weeks
  The results are presented as reaching or not reaching 150 minutes of moderate physical activity per week.
The person's own goals regarding function collected with the Patient Specific Functional Scale (PSFS). | At baseline, and post-intervention/after 12 weeks
  The participant will choose three activities of individual importance and rate the ability to perform each activity on a scale from 0 (not able to perform the activity) to 10 (can perform the activity unhindered).
Health related quality of life collected with the EuroQol five dimension scale (EQ-5D 3L). | At baseline, and post-intervention/after 12 weeks
  Reported as an index utility score between 0 to 1 (a higher score indicates better health state) and a visual analogue scale of self-related overall health ranging from 0 to 100 (a higher score indicates better overall health).
Self-reported disability collected with the Oswestry Disability Index (ODI). | At baseline, and post-intervention/after 12 weeks
  Score range from 0 to 50. Higher scores represent greater disability.
Depressed mood collected with the depression subscale of the Hospital Anxiety and Depression Scale. | At baseline, and post-intervention/after 12 weeks
  Score range from 0 to 21. A score of 8 or more indicated depression.
Pain intensity level in the leg and back reported with the Numeric Rating Scale (NRS). | At baseline, and post-intervention/after 12 weeks
  On a scale from 0 to 10, where a higher reported number means higher pain intensity.
Catastrophizing thoughts related to pain collected with the Pain Catastrophizing Scale (PCS). | At baseline, and post-intervention/after 12 weeks
  Score range from 0 to 52. Higher scores mean higher degree of catastrophizing thoughts related to pain.
Patient-reported kinesiophobia collected with the Swedish version of the Tampa Scale of Kinesiophobia (TSK-SV). | At baseline, and post-intervention/after 12 weeks
  Score range from 17 to 68. Higher scores mean higher degree of fear of movement.
General self-efficacy collected with the General Self-efficacy Scale (GSE). | At baseline, and post-intervention/after 12 weeks
  Score range from 10 to 40. Higher scores mean higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Mari K Lundberg, Principal Investigator — Sophiahemmet Högskola
Locations (2):
- Sweden (2):
  - Capio Spine Center Göteborg, Västra Frölunda, Gothenburg
  - Ryggkirurgiskt centrum Stockholm, Stockholm, Stockholm County

IPD SHARING:
Plan to Share IPD: No
The data in the study will be pseudonymised (coded) personal data, and Swedish legislation prohibits us from sharing this completely open. The dataset will only include data from 30 human research participants. Due to the small sample size risk of identification of individual participants exists even though data is coded. Some data is available upon request, which will be handled according to the relevant legislation.

REFERENCES:
- [Derived] Karlsson E, Hanafi R, Brisby H, Fors A, Kemani M, Hedman H, Nijs J, Lundberg M. Get Back, a person-centred digital programme targeting physical activity for patients undergoing spinal stenosis surgery-a study protocol of a randomized feasibility study. Pilot Feasibility Stud. 2024 Jan 26;10(1):16. doi: 10.1186/s40814-023-01433-9. PMID 38279131